CLINICAL TRIAL: NCT06441175
Title: Comparison of the Effectiveness of Cricoid Pressure on Upper Esophageal Obstruction During Videolaryngoscopy Versus Direct Laryngoscopy: a Randomized, Crossover Study
Brief Title: Effectiveness of Cricoid Pressure During Videolaryngoscopy Versus Direct Laryngoscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CP during videolaryngoscopy
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Cricoid Pressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-V group (Experimental): the group that performs direct laryngoscopy first and then videolaryngoscopy
  Interventions: Other: Intubation device order
- V-D group (Experimental): the group that performs videolaryngoscopy first and then directlaryngoscopy
  Interventions: Other: Intubation device order

INTERVENTIONS:
Other: Intubation device order — D-V group: the group that performs direct laryngoscopy first and then videolaryngoscopy.
  V-D group: the group that performs video laryngoscopy first and then directlaryngoscopy."

SUMMARY:
Compare the success rate of upper esophageal obstruction with cricoid pressure during videolaryngoscopy and direct laryngoscopy.

DETAILED DESCRIPTION:
Even with appropriate cricoid pressure, the lifting force of the laryngoscope during direct laryngoscopy for tracheal intubation may counteract the cricoid pressure, making esophageal obstruction ineffective. Compared to direct laryngoscopy, videolaryngoscopy requires less lifting force, and thus, the success rate of esophageal obstruction may be higher. This study aims to compare the success rate of upper esophageal obstruction with cricoid pressure during videolaryngoscopy and direct laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled to have general anesthesia with tracheal intubation

Exclusion Criteria:

* Gastroesophageal reflux disease, achalasia, bowel obstruction,
* BMI > 35 kg/m2
* Uncontrolled diabetes
* Pregnancy
* Previous esophageal, and gastric surgery
* Dental damage or anticipated difficult airways
* Who do not consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of esophageal obstruction during cricoid pressure | During general anesthesia induction
  Success rate of esophageal obstruction during cricoid pressure

SECONDARY OUTCOMES:
Esophageal diameter | During cricoid pressure
  Esophageal diameter measured by ultrasound
percentage of glottic opening score | During cricoid pressure
  percentage of glottic opening
Cormack-Lehane grade | During cricoid pressure
  views obtained by laryngoscopy

CONTACTS AND LOCATIONS:
Overall Officials: TAE KYONG KIM, Principal Investigator — SMG-SNU Boramae Medical Center